CLINICAL TRIAL: NCT02409459
Title: A Blinded, Randomized, Placebo-Controlled Study to Investigate the Efficacy and Safety of Injectafer (Ferric Carboxymaltose) in the Treatment of Iron Deficient Patients With Fibromyalgia
Brief Title: Blinded Randomized Placebo-Controlled Study Efficacy and Safety of Injectafer in ID Patients With Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1VIT14038
Record Dates: First submitted 2015-04-01; First posted 2015-04-06 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-01

CONDITIONS: Iron Deficiency; Fibromyalgia
MeSH Terms: conditions — Iron Deficiencies; Fibromyalgia | interventions — ferric carboxymaltose; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Injectafer (Experimental): 15 mg/kg up to 750 mg undiluted blinded dose of IV Injectafer (ferric carboxymaltose) at 100 mg/minute
  Interventions: Drug: Injectafer
- Placebo (Placebo Comparator): 15 cc of Normal Saline IV push at 2 ml/minute
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Injectafer
  Other Names: Ferric Carboxymaltose (FCM)
  Arms: Injectafer
Drug: Placebo — Normal saline solution
  Other Names: Saline solution
  Arms: Placebo

SUMMARY:
This study investigates the efficacy and safety of an IV iron Injectafer in the treatment of iron deficient patients with fibromyalgia. Eligible subjects will be randomized in a 1:1 ratio to receive Injectafer or Placebo on days 0 and 5. All treated subjects will be followed for efficacy and safety for 42 days.

DETAILED DESCRIPTION:
This is a blinded, randomized, placebo-controlled study. All subjects who meet the inclusion requirements and no exclusion criteria will be entered into an up to 14 day screening phase. Eligible subjects will be randomized in a 1:1 ratio to receive Injectafer or Placebo on days 0 and 5. All treated subjects will be followed for efficacy and safety for 42 days. Subjects will visit the clinic on days 0 and 5 for treatment, and then on days 14, 28, and 42. The subject's participation in the study will be for approximately 42 days from day 0.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject's ≥ 18 years of age, able to give informed consent to the study.
* Fibromyalgia diagnosis based on The 2011 modification of the American College of Rheumatology (ACR) 's 2010 preliminary criteria for diagnosing fibromyalgia (2011ModCr)
* A baseline score ≥ 60 on the FIQR
* Subject's current medications to treat fibromyalgia, including pain medicines, anti-depressants, sleep medications must be on a stable dose for at least 30 days.
* Subject's current narcotic medication must be on a stable dose for at least 30 days prior to randomization
* Subjects at risk for pregnancy must have a negative pregnancy test at baseline and be practicing an acceptable form of birth control: have had a hysterectomy or tubal ligation, or otherwise be incapable of pregnancy, or have practiced any of the following methods of contraception for at least one month prior to study entry: hormonal contraceptives, spermicide and barrier, intrauterine device, partner sterility.

Exclusion Criteria:

* Parenteral iron use within 4 weeks prior to screening.
* History of > 10 blood transfusions in the past 2 years.
* Anticipated need for blood transfusion during the study.
* Known hypersensitivity reaction to any component of Injectafer® (Ferric Carboxymaltose).
* Current or acute or chronic infection other than viral upper respiratory tract infection
* Malignancy (other than basal or squamous cell skin cancer or the subject has been cancer free for ≥ 5 years).
* Active inflammatory arthritis (e.g. rheumatoid arthritis, SLE).
* Pregnant or lactating women.
* Severe peripheral vascular disease with significant skin changes.
* Seizure disorder currently being treated with medication.
* Baseline ferritin ≥ 50 ng/mL.
* Baseline TSAT ≥ 20%.
* History of hemochromatosis or hemosiderosis or other iron storage disorders.
* Known positive hepatitis with evidence of active disease.
* Hemoglobin greater than the upper limit of normal.
* Calcium or phosphorous outside the normal range.
* Known positive hepatitis B antigen (HBsAg) or hepatitis C viral antibody (HCV) with evidence of active hepatitis (i.e., AST/ALT greater than the upper limit of normal).
* Known positive HIV-1/HIV-2 antibodies (anti-HIV)
* Received an investigational drug within 30 days before randomization.
* Chronic alcohol or drug abuse within the past 6 months.
* Any other pre-existing laboratory abnormality, medical condition or disease which in view of the investigator participation in this study may put the subject at risk.
* Subject unable to comply with the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Falone, MD, Study Director — American Regent, Inc.
Locations (1):
- Clinical Research Solutions, Franklin, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Boomershine CS, Koch TA, Morris D. A Blinded, Randomized, Placebo-Controlled Study to Investigate the Efficacy and Safety of Ferric Carboxymaltose in Iron-Deficient Patients with Fibromyalgia. Rheumatol Ther. 2018 Jun;5(1):271-281. doi: 10.1007/s40744-017-0088-9. Epub 2017 Nov 17. PMID 29149437

RESULTS

PARTICIPANT FLOW:
Groups:
- Injectafer: 15 mg/kg up to 750 mg undiluted blinded dose of IV Injectafer (ferric carboxymaltose) at 100 mg/minute
  Injectafer
- Placebo: 15 cc of Normal Saline IV push at 2 ml/minute
  Normal Saline
Period: Overall Study
Arm/Group | Injectafer | Placebo
Started | 41 | 40
Completed | 40 | 39
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Group B: Placebo
- Injectafer: Group A: Injectafer
- Total: Total of all reporting groups
Arm/Group | Placebo | Injectafer | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (10.85) | 41 (11.07) | 43 (10.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African American | 7 | 7 | 14
  Race: Asian | 0 | 1 | 1
  Race: Caucasian | 30 | 33 | 63
  Race: Hispanic | 2 | 0 | 2
  Race: Other | 1 | 0 | 1
History of iron intolerance [Count of Participants; unit: Participants]
  No | 37 | 35 | 72
  Yes | 3 | 6 | 9
History of drug allergy [Count of Participants; unit: Participants]
  No | 17 | 21 | 38
  Yes | 23 | 20 | 43
IRLS score per Arm/Group [Mean (Standard Deviation); unit: units on a scale] — 'International Restless Legs Syndrome Study Group Rating Scale' (IRLS) The IRLS is composed of 10 items. It gives a global score for all 10 items that is most commonly used as an overall severity score. 9 of the 10 items investigate two dimensions of the RLS severity. Item 3 is part of the diagnostic criteria and does not belong to any of the two dimensions. It is used for the total score for overall RLS severity.
  Symptom severity subscale: 0-24 Impact on daily living subscale: 0-12 Global score: 0-40 For all scores, higher score = higher symptom impact.
  units on a scale | 16.3 (14.9) | 13.4 (13.16) | 14.8 (14.04)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With a ≥13 Point Improvement in FIQR Score
Description: The primary efficacy endpoint was the percentage of subjects who had a ≥13-point improvement in the FIQR from baseline to Day 42.
Time Frame: Day 42
Population: The Safety population consisted of all subjects who received at least one dose of randomized treatment. The Efficacy Evaluable Population consisted of all subjects who received at least 1 dose of randomized treatment with at least 1 completed post treatment FIQR evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Injectafer | Placebo
Number analyzed (Participants) | 39 | 39
Participants | 30 | 26

2. Secondary Outcome: Change in BPI, Pain Interference
Description: The short version of the Brief Pain Inventory (BPI) includes front and back body diagrams, 4 pain severity items and 7 pain interference items rated on 0-10 scales (with 0 being the best outcome and 10 being the worst outcome), and a question about percentage of pain relief by analgesics. The Pain Interference Score is calculated by adding the scores for the 7 pain interference questions and then dividing by 7 to give a score out of 10.
Time Frame: Change from Baseline in Brief Pain Inventory Pain Interference Score at Day 42
Population: Patients without a particular measure at a required time point were excluded from the analysis of that measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Injectafer | Placebo
Number analyzed (Participants) | 38 | 39
units on a scale | -4.1 (3.3) | -2.3 (2.6)

3. Secondary Outcome: Change in FIQR Score
Description: The FIQR has 21 individual questions. All questions are based on an 11-point numeric rating scale of 0 to 10, with 10 being 'worst' and all questions are framed in the context of the past 7 days. The summed score for function (range 0 to 90) is divided by 3, the summed score for overall impact (range 0 to 20) is not changed, and the summed score for symptoms (range 0 to 100) is divided by 2. The total FIQR is the sum of the three modified domain scores.
Time Frame: Change from Baseline in FIQR score at Day 42
Population: Patients without a particular measure at a required time point were excluded from the analysis of that measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Injectafer | Placebo
Number analyzed (Participants) | 38 | 39
units on a scale | -45.0 (29.5) | -29.7 (27.0)

4. Secondary Outcome: Change in BPI, Pain Severity
Description: The short version of the Brief Pain Inventory (BPI) includes front and back body diagrams, 4 pain severity items and 7 pain interference items rated on 0-10 scales (with 0 being the best outcome and 10 being the worst outcome), and a question about percentage of pain relief by analgesics. The Pain Severity Score is calculated by adding the scores for the 4 pain severity questions and then dividing by 4 to give a severity score out of 10.
Time Frame: Change from Baseline in Brief Pain Inventory Pain Severity Score at Day 42
Population: Patients without a particular measure at a required time point were excluded from the analysis of that measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Injectafer | Placebo
Number analyzed (Participants) | 38 | 39
units on a scale | -3.1 (2.7) | -1.8 (2.1)

5. Secondary Outcome: Change in Fatigue Visual Numeric Scale
Description: Scores range from 0 to 10, with the higher score indicating more fatigue.
Time Frame: Change from Baseline in Fatigue Visual Numeric Scale at Day 42
Population: Patients without a particular measure at a required time point were excluded from the analysis of that measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Injectafer | Placebo
Number analyzed (Participants) | 37 | 39
units on a scale | -3.7 (3.2) | -1.7 (2.2)

6. Secondary Outcome: Change in Iron Indices, Serum Ferritin
Time Frame: Change from Baseline in Iron Indices, Serum ferritin at Day 42
Population: Patients without a particular measure at a required time point were excluded from the analysis of that measure.
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Injectafer | Placebo
Number analyzed (Participants) | 39 | 38
ug/L | 292.5 (145.9) | 2.0 (13.8)

7. Secondary Outcome: Change in Iron Indices - Transferrin Saturation
Time Frame: Change from baseline in Iron Indices, Transferrin saturation, at Day 42
Population: Patients without a particular measure at a required time point were excluded from the analysis of that measure.
Measure: Mean (Standard Deviation); unit: percent of transferrin saturation
Arm/Group | Injectafer | Placebo
Number analyzed (Participants) | 39 | 38
percent of transferrin saturation | 24.4 (11.4) | 5.8 (15.1)

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Injectafer | Placebo
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/40
Other Adverse Events (participants affected / at risk) | 16/41 | 2/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Injectafer (N=41) | Placebo (N=40)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 6 (6) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No